CLINICAL TRIAL: NCT00496470
Title: A 12-week, Double-blind, Randomised, Parallel Group, Multi-centre, Study to Evaluate Efficacy and Safety of Budesonide/Formoterol (Symbicort Turbuhaler®) 320/9 µg One Inhalation Twice Daily on Top of Tiotropium (Spiriva®) 18 µg One Inhalation Once Daily
Brief Title: Evaluation of Efficacy and Safety of Symbicort® as an add-on Treatment to Spiriva® in Patients With Severe COPD.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5892C00015; Eudract no:2006-006796-21
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Results first posted 2012-11-09 (Estimated); Last update posted 2012-11-09 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Obstructive Pulmonary Disease, COPD
Keywords: Chronic Obstructive Pulmonary Disease, COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide, Formoterol Fumarate Drug Combination; Budesonide; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Symbicort+TIO (Active Comparator): Symbicort Turbuhaler® (budesonide/formoterol) 320/9 mcg, one inhalation twice daily and Spiriva® (tiotropium) 18 mcg, one inhalation once daily
  Interventions: Drug: Symbicort (budesonide/formoterol turbuhaler 320/9ug)
- Spiriva® + Placebo Turbuhaler (Active Comparator): Spiriva® (tiotropium) 18 mcg, one inhalation once daily and placebo Turbuhaler one inhalation once daily
  Interventions: Drug: Spiriva (tiotropium bromide 18ug)

INTERVENTIONS:
Drug: Symbicort (budesonide/formoterol turbuhaler 320/9ug) — Symbicort (budesonide/formoterol turbuhaler 320/9ug)
  Arms: Symbicort+TIO
Drug: Spiriva (tiotropium bromide 18ug) — Spiriva (tiotropium bromide 18ug)
  Arms: Spiriva® + Placebo Turbuhaler

SUMMARY:
The purpose of this study is to investigate the effect of combined treatment with Symbicort and Spiriva, in terms of improvement of lung function, symptoms and inflammatory markers, in patients with severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* >=40 years of age, diagnosed COPD with symptoms >=2 years, pre-bronchodilatory FEV1 <=50% of PN

Exclusion Criteria:

* Current respiratory tract disorder other than COPD, history of asthma or rhinitis, significant or unstable cardiovascular disorder

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2007-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Andersson, MD, Study Director — AstraZeneca R&D Lund; Tobias Welte, MD, Principal Investigator — Hannover Medical School
Locations (93):
- Australia (10):
  - Research Site, Concord, New South Wales
  - Research Site, Sydney, New South Wales
  - Research Site, Auchenflower, Queensland
  - Research Site, Carina Heights, Queensland
  - Research Site, North Mackay, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Daw Park, South Australia
  - Research Site, Clayton, Victoria
  - Research Site, Malvern, Victoria
  - Research Site, Nedlands, Western Australia
- Canada (11):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Mississauga, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, La Malbaie, Quebec
  - Research Site, Trois-rivires, Quebec
  - Research Site, Saskatoon, Saskatchewan
  - Research Site, Québec
- France (14):
  - Research Site, Chamalières
  - Research Site, Creil
  - Research Site, Férolles-Attilly
  - Research Site, Grasse
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Metz
  - Research Site, Montpellier
  - Research Site, Perpignan
  - Research Site, Poitiers
  - Research Site, Saint-Laurent-du-Var
  - Research Site, Sélestat
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (9):
  - Research Site, Berlin
  - Research Site, Gelsenkirchen
  - Research Site, Hagen
  - Research Site, Hanover
  - Research Site, Kassel
  - Research Site, Koblenz
  - Research Site, Leipzig
  - Research Site, Marburg
  - Research Site, Potsdam
- Hungary (12):
  - Research Site, Aszód
  - Research Site, Baja
  - Research Site, Balassagyarmat
  - Research Site, Budapest
  - Research Site, Cegléd
  - Research Site, Debrecen
  - Research Site, Füzesabony
  - Research Site, Jászberény
  - Research Site, Komló
  - Research Site, Nyíregyháza
  - Research Site, Törökbálint
  - Research Site, Vásárosnamény
- Poland (9):
  - Research Site, Bydgoszcz
  - Research Site, Chrzanów
  - Research Site, Iława
  - Research Site, Krakow
  - Research Site, Piekary Śląskie
  - Research Site, Tarnów
  - Research Site, Turek
  - Research Site, Zawadzkie
  - Research Site, Łomża
- Slovakia (13):
  - Research Site, Košice
  - Research Site, Liptovský Hrádok
  - Research Site, Lučenec
  - Research Site, Nové Mesto nad Váhom
  - Research Site, Nové Zámky
  - Research Site, Piešťany
  - Research Site, Poprad
  - Research Site, Považská Bystrica
  - Research Site, Prešov
  - Research Site, Prievidza
  - Research Site, Revúca
  - Research Site, Trnava
  - Research Site, Žilina
- Spain (6):
  - Research Site, Barcelona, Catalonia
  - Research Site, Reus (tarragona), Catalonia
  - Research Site, Pontevedra, Galicia
  - Research Site, Madrid, Madrid
  - Research Site, Requena (valencia), Valencia
  - Research Site, Valencia, Valencia
- Sweden (9):
  - Research Site, Åtvidaberg
  - Research Site, Höllviken
  - Research Site, Limhamn
  - Research Site, Lund
  - Research Site, Malmo
  - Research Site, Motala
  - Research Site, Stockholm
  - Research Site, Uppsala
  - Research Site, Lindesberg, Örebro County

REFERENCES:
- [Derived] Nielsen R, Kankaanranta H, Bjermer L, Lange P, Arnetorp S, Hedegaard M, Stenling A, Mittmann N. Cost effectiveness of adding budesonide/formoterol to tiotropium in COPD in four Nordic countries. Respir Med. 2013 Nov;107(11):1709-21. doi: 10.1016/j.rmed.2013.06.007. Epub 2013 Jul 13. PMID 23856511
- [Derived] Mittmann N, Hernandez P, Mellstrom C, Brannman L, Welte T. Cost effectiveness of budesonide/formoterol added to tiotropium bromide versus placebo added to tiotropium bromide in patients with chronic obstructive pulmonary disease: Australian, Canadian and Swedish healthcare perspectives. Pharmacoeconomics. 2011 May;29(5):403-14. doi: 10.2165/11590380-000000000-00000. PMID 21504240
- [Derived] Partridge MR, Miravitlles M, Stahl E, Karlsson N, Svensson K, Welte T. Development and validation of the Capacity of Daily Living during the Morning questionnaire and the Global Chest Symptoms Questionnaire in COPD. Eur Respir J. 2010 Jul;36(1):96-104. doi: 10.1183/09031936.00123709. Epub 2009 Nov 6. PMID 19897551
- [Derived] Welte T, Miravitlles M, Hernandez P, Eriksson G, Peterson S, Polanowski T, Kessler R. Efficacy and tolerability of budesonide/formoterol added to tiotropium in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2009 Oct 15;180(8):741-50. doi: 10.1164/rccm.200904-0492OC. Epub 2009 Jul 30. PMID 19644045

RESULTS

PARTICIPANT FLOW:
Groups:
- Symbicort+Tiotropium: Symbicort Turbuhaler® (budesonide/formoterol) 320/9 mcg, one inhalation twice daily and Spiriva® (tiotropium) 18 mcg, one inhalation once daily
- Placebo+Tiotropium: Spiriva® (tiotropium) 18 mcg, one inhalation once daily and placebo Turbuhaler one inhalation once daily
Period: Overall Study
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Started | 329 | 331
Received Study Medication | 329 | 330
Completed | 303 | 302
Not Completed | 26 | 29
Not completed — Adverse Event | 8 | 10
Not completed — Withdrawal by Subject | 5 | 12
Not completed — Incorrectly enrolled | 13 | 5
Not completed — Other reason | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium | Total
Number analyzed (Participants) | 329 | 331 | 660
Age Continuous [Mean (Full Range); unit: Years] | 62.4 [40 to 85] | 62.5 [41 to 82] | 62.45 [40 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 86 | 164
  Male | 251 | 245 | 496

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Pre-dose
Description: Change in the pre-dose FEV1from baseline to week 12 (calculated as a mean using all available data of treatment period between week 1 and week 12)
Time Frame: Baseline to 12 weeks
Population: Full analysis set (FAS) was performed and was based on data from all subjects who were randomized, took at least 1 dose of study medication, and contributed sufficient data for calculation of this outcome Measure.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 323 | 327
Liters | 0.064 (0.198) | -0.001 (0.168)

2. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 5 Min Post-dose
Description: Change in the 5 min post-dose FEV1from baseline to week 12 (calculated as a mean using all available data of treatment period between week 1 and week 12)
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 329 | 330
Liters | 0.165 (0.184) | 0.042 (0.14)

3. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) 60 Min Post-dose
Description: Change in the 60 min post-dose FEV1from baseline to week 12 (calculated as a mean using all available data of treatment period between week 1 and week 12)
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 329 | 330
Liters | 0.214 (0.209) | 0.083 (0.157)

4. Secondary Outcome: Forced Vital Capacity (FVC) Pre-dose
Description: Change in the pre-dose FVC from baseline to week 12 (calculated as a mean using all available data of treatment period between week 1 and week 12)
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 323 | 327
Liters | 0.07 (0.341) | 0.014 (0.348)

5. Secondary Outcome: Forced Vital Capacity (FVC) 5 Minutes Post-dose
Description: Change in the 5 min post-dose FVC from baseline to week 12 (calculated as a mean using all available data of treatment period between week 1 and week 12)
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 329 | 330
Liters | 0.266 (0.32) | 0.106 (0.296)

6. Secondary Outcome: Forced Vital Capacity (FVC) 60 Minutes Post-dose
Description: Change in the 60 min post-dose FVC from baseline to week 12 (calculated as a mean using all available data of treatment period between week 1 and week 12
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 329 | 330
Liters | 0.353 (0.357) | 0.19 (0.319)

7. Secondary Outcome: Inspiratory Capacity (IC) Pre-dose
Description: Change in the pre-dose IC from baseline to week 12 (calculated as a mean using all available data of treatment period between week 1 and week 12)
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 314 | 309
Liters | 0.078 (0.35) | 0.014 (0.389)

8. Secondary Outcome: Inspiratory Capacity (IC) 60 Minutes Post-dose
Description: Change in the 60 min post-dose IC from baseline to week 12 (calculated as a mean using all available data of treatment period between week 1 and week 12)
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 318 | 310
Liters | 0.26 (0.353) | 0.149 (0.359)

9. Secondary Outcome: St George's Respiratory Questionnaire for COPD Patients (SGRQ-C) Score
Description: Change in total score from baseline (Visit 3) to end of treatment (Visit 6, or last available visit).
  SGRQ-C is a health related quality of life questionnaire consisting of 40 items divided into two components: 1) symptoms, 2) activity& impacts. The lowest possible value is zero and the highest 100. Higher values correspond to greater impairment in quality of life.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 315 | 320
Score on a scale | -4.12 (12.81) | -1.99 (12.77)

10. Secondary Outcome: Morning Peak Expiratory Flow (PEF) Pre-dose
Description: Daily diary record. Change in average values from run-in to the full treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 329 | 330
Liters/minute | 5.12 (38.3) | -3.52 (24.7)

11. Secondary Outcome: Evening Peak Expiratory Flow (PEF) Pre-dose
Description: Daily diary record. Change in average values from run-in to the full treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 329 | 329
Liters/minute | 2.82 (37.6) | -5.54 (28.9)

12. Secondary Outcome: Morning Peak Expiratory Flow (PEF) 5 Min Post-dose
Description: Daily diary record. Change in average values from run-in to the full treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 294 | 307
Liters/minute | 16.71 (42.6) | 1.1 (26.5)

13. Secondary Outcome: Morning Peak Expiratory Flow (PEF) 15 Min Post-dose
Description: Daily diary record. Change in average values from run-in to the full treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 293 | 311
Liters/minute | 20.4 (43.7) | 5.2 (28.3)

14. Secondary Outcome: Morning Diary FEV1 Pre-dose
Description: Daily diary record. Change in average values from run-in to the full treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 219 | 233
Liters | 0.054 (0.201) | -0.046 (0.185)

15. Secondary Outcome: Evening Diary FEV1, Pre-dose
Description: Daily diary record. Change in average values from run-in to the full treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 221 | 237
Liters | 0.012 (0.223) | -0.065 (0.249)

16. Secondary Outcome: Morning Diary FEV1, 5 Minutes Post-dose
Description: Daily diary record. Change in average values from run-in to the full treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 191 | 205
Liters | 0.169 (0.224) | -0.018 (0.189)

17. Secondary Outcome: Morning Diary FEV1, 15 Minutes Post-dose
Description: Daily diary record. Change in average values from run-in to the full treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 190 | 208
Liters | 0.209 (0.236) | 0.014 (0.201)

18. Secondary Outcome: Global Chest Symptoms Questionnaire (GCSQ) Score, Pre-dose
Description: Daily diary record. Change in average values from run-in to the full treatment period.
  The GCSQ consisted of two questions that required the patient to rate shortness of breath and feelings of chest tightness. The patients recorded their response on a five-point Likert-type scale ranging from 0 (not at all) to 4 (extremely), the total score being calculated as the average score of the two questions.
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 329 | 328
Scores on a scale | -0.143 (0.453) | -0.006 (0.438)

19. Secondary Outcome: GCSQ Score, 5 Minutes Post-dose
Description: as for outcome 18
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 296 | 305
Scores on a scale | -0.325 (0.508) | -0.202 (0.46)

20. Secondary Outcome: GCSQ Score, 15 Minutes Post-dose
Description: as for outcome 18
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 293 | 309
Scores on a scale | -0.404 (-0.526) | -0.28 (-0.501)

21. Secondary Outcome: Capacity of Day Living in the Morning (CDLM) Score
Description: Daily diary record. Change in average values from run-in to the full treatment period.
  The CDLM questionnaire is as a questionnaire to report on patient's ability to carry out each of six different morning activities (score ranging from 0 "not performed" to 1"performed") and rank the difficulty of performing each of those activities (score ranging from 0 "so difficult that the activity could not be carried out by the patient on their own" to 5 "activity was not at all difficult to carry out". Total score for each morning activity range from 0-6. Total score for whole CDLM questionnaire range from 0-36.
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 281 | 294
Scores on a scale | 0.202 (0.467) | 0.07 (0.435)

22. Secondary Outcome: Use of Rescue Medication, Night
Description: Daily diary record - Night, after evening measurement till morning. Change in average values from run-in to the full treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Inhalations
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 329 | 330
Inhalations | -0.279 (0.7) | 0.022 (0.743)

23. Secondary Outcome: Use of Rescue Medication, Morning
Description: Daily diary record - Morning, after morning measurement till midday. Change in average values from run-in to the full treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Inhalations
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 281 | 294
Inhalations | -0.417 (0.758) | -0.124 (0.877)

24. Secondary Outcome: Use of Rescue Medication, Day
Description: Daily diary record - Day, after morning measurement till evening. Change in average values from run-in to the full treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Inhalations
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 329 | 329
Inhalations | -0.745 (1.286) | -0.371 (1.622)

25. Secondary Outcome: Use of Rescue Medication, Total
Description: Daily diary record - Total, 24 hours, during the night, and during the day. Change in average values from run-in to the full treatment period
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Inhalations
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 329 | 329
Inhalations | -1.024 (1.704) | -0.347 (2.102)

26. Secondary Outcome: COPD Symptoms, Breathing Score
Description: Daily diary record. Change in average values from run-in to the full treatment period. Symptom scale 0 - 4 (0) None (1) Mild (2) Moderate (3) Marked (4) Severe
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 329 | 329
Units on a Scale | -0.177 (0.503) | -0.049 (0.5)

27. Secondary Outcome: COPD Symptoms, Sleeping Score
Description: as for outcome 26
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 329 | 330
Units on a Scale | -0.197 (0.45) | -0.045 (0.462)

28. Secondary Outcome: COPD Symptoms, Chest Score
Description: as for outcome 26
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 329 | 329
Units on a Scale | -0.184 (0.5) | -0.061 (0.473)

29. Secondary Outcome: COPD Symptoms, Cough Score
Description: as for outcome 26
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 329 | 329
Units on a Scale | -0.246 (0.567) | -0.079 (0.545)

30. Secondary Outcome: Severe COPD Exacerbations
Description: Patients with worsening of COPD leading to treatment with systemic steroids (oral or parenteral), emergency room treatment or hospitalisation
Time Frame: 12 weeks
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 329 | 330
Participants | 25 | 61

31. Secondary Outcome: Serum High-sensitivity C-reactive Protein (hsCRP)
Description: Ratio of treatment period mean to run-in value
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 304 | 309
Ratio | 0.91 [0.5 to 1.76] | 0.97 [0.6 to 1.54]

32. Secondary Outcome: Serum Interleukin 6 (IL-6)
Description: Ratio of treatment period mean to run-in value
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 304 | 309
Ratio | 1.0 [0.72 to 1.56] | 1.0 [0.67 to 1.56]

33. Secondary Outcome: Serum Interleukin 8 (IL-8)
Description: Ratio of treatment period mean to run-in value
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 304 | 309
Ratio | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]

34. Secondary Outcome: Serum Monocyte Chemoattractant Protein-1 (MCP-1)
Description: Ratio of treatment period mean to run-in value
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 304 | 309
Ratio | 0.95 [0.78 to 1.15] | 0.95 [0.79 to 1.11]

35. Secondary Outcome: Serum Soluble Tumor Necrosis Factor-alpha (sTNF-alpha)
Description: Ratio of treatment period mean to run-in value
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 304 | 309
Ratio | 0.97 [0.85 to 1.08] | 0.98 [0.88 to 1.1]

36. Secondary Outcome: Serum Tumor Necrosis Factor-alpha (TNF-alpha)
Description: Ratio of treatment period mean to run-in value
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 304 | 309
Ratio | 1.0 [0.69 to 1.28] | 1.0 [0.67 to 1.2]

37. Secondary Outcome: Serum Vascular Cell Adhesion Molecule-1 (VCAM-1)
Description: Ratio of treatment period mean to run-in value
Time Frame: Baseline to 12 weeks
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Ratio
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Number analyzed (Participants) | 304 | 309
Ratio | 0.96 [0.87 to 1.06] | 0.99 [0.91 to 1.09]

ADVERSE EVENTS:
Arm/Group | Symbicort+Tiotropium | Placebo+Tiotropium
Serious Adverse Events (participants affected / at risk) | 10/329 | 16/330
Other Adverse Events (participants affected / at risk) | 0/329 | 0/330
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort+Tiotropium (N=329) | Placebo+Tiotropium (N=330)
Acute Coronary Syndrome (Cardiac disorders) | 1 | 0
Atrioventricular Block Second Degree (Cardiac disorders) | 0 | 1
Infective Exacerbation of Chronic Obstructive Airways Disease (Infections and infestations) | 2 | 2
Pneomonia (Infections and infestations) | 1 | 1
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 1
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to any publication or disclosure, the PI provides AstraZeneca with preliminary data and drafts and with the proposed final manuscript. AstraZeneca shall have a period of 30 days from receipt of the proposed final manuscript to review it and may within such time frame require that submission for publication or disclosure be delayed.